CLINICAL TRIAL: NCT04398069
Title: Hemodynamic Optimisation Guided With Transcranial Doppler in Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor head of the anesthesia and intensive care department, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Hemodynamic optimization ICU
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Trans Cranial Doppler Ultrasonography in Heamodynamic Optimisation in Septic Shock
Keywords: Trans cranial doppler ultrasonography, hemodynamics, septic shock, sepsis associated encephalopathy
MeSH Terms: conditions — Shock, Septic; Sepsis-Associated Encephalopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Group (No Intervention): standard hemodynamic goals and catecholamin infusion to achieve: mean arterial pressure > or equal to 65 mmHg and diastolic arterial pressure > ou equal to 50 mmHg within the first 60 minutes.
- personalized hemodynamic goals Group (Experimental): Personalized hemodynamic goals and catecholamin infusion to achieve normal cerebral perfusion assessed by transcranial doppler: PI < 1,2.
  Interventions: Procedure: hemodynamic optimisation aiming to achieve normal cerebral perfusion

INTERVENTIONS:
Procedure: hemodynamic optimisation aiming to achieve normal cerebral perfusion — hemodynamic optimisation aiming to achieve normal cerebral perfusion: titration of catecholamin infusion.
  Arms: personalized hemodynamic goals Group

SUMMARY:
Randomized, controlled, prospective trial, including ICU patients with Sepsis or septic Shock, at the early phase.

patients will be randomized in 2 groups regarding the hemodynamic management and catecholamin doses:

* Group 1: standard hemodynamic goals and catecholamin infusion to achieve: mean arterial pressure > or equal to 65 mmHg and diastolic arterial pressure > ou equal to 50 mmHg within the first 60 minutes.
* Group 2: personalized hemodynamic goals and catecholamin infusion until normal transcranial doppler: IP<1,2.

DETAILED DESCRIPTION:
Randomized, controlled, prospective trial, including ICU patients with Sepsis or septic Shock, at the early phase.

patients will be randomized in 2 groups regarding the hemodynamic management and catecholamin doses:

* Group 1: standard hemodynamic goals and cathecolamin infusion to achieve: mean arterial pressure > or equal to 65 mmHg and diastolic arterial pressure > ou equal to 50 mmHg within the first 60 minutes.
* Group 2: personalized hemodynamic goals and cathecolamin infusion until normal transcranial doppler: IP<1,2.

For the 2 groups, standard management including: microbiological sampling, early broad spectrum anti infective therapy, fluid management and decreasing of blood lactate levels, will be aimed within the first 60 minutes.

For the Group 2 patients: personalized hemodynamic management will be maintained during 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* All ICU patients presenting septic shock
* No criteria of traumatic or vascular brain injury

Exclusion Criteria:

* Patients with refractory septick shock
* rapid fatal evolution: before 72 hours
* No individualisation of the MCA ultrasonographic window

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
mortality at day 28 | 28 days after ICU admission
  Mortality at day 28

SECONDARY OUTCOMES:
Incidence of sepsis associated encephalopathy | 28 days after ICU admission
  sepsis associated encephalopathy assessed by CAM-ICU and GCS scores
Incidence of sepsis related organ failures | 28 days after ICU admission
  sepsis related organ failures assessed with SOFA score
Length of ICU stay | 30 days after end of randomization
  Length of ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Mhamed Sami Mebazaa, Professor, Principal Investigator — Mongi Slim Hospital
Locations (1):
- Mongi Slim Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No